CLINICAL TRIAL: NCT03386760
Title: Evaluation of an Ultra-speed Picosecond Laser for Treating Tattoos
Acronym: PicoS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-PP-07
Record Dates: First submitted 2017-12-18; First posted 2017-12-29 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Tattoo; Pigmentation
Keywords: tattoo

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A- Ultra-Speed Picosecond laser (Experimental): Utilisation of Ultra-speed Picosecond laser for tattoo depigmentation
  Interventions: Device: Laser Utilisation PicoSecond
- B- Nanosecond laser (Active Comparator): Utilisation of Nanosecond laser for tattoo depigmentation
  Interventions: Device: Laser Utilisation Nano-second

INTERVENTIONS:
Device: Laser Utilisation PicoSecond — Laser utilisation for tattoo depigmentation
  1 session every month for a total of 3 sessions
  Arms: A- Ultra-Speed Picosecond laser
Device: Laser Utilisation Nano-second — Laser utilisation for tattoo depigmentation
  1 session every month for a total of 3 sessions
  Arms: B- Nanosecond laser

SUMMARY:
The investigators developed an ultra-speed picosecond laser (20ps) with a 20gHz repetition rate that provide very promising results in vitro and in ex vivo skin to remove skin tattoos.

The aim of this study is to evaluate the efficacy and tolerance of a new ultra-speed picosecond laser and to compare it to a nanosecond laser for treating black tattoos.

In a first phase of the study 10 patients with black tattoos will be treated with increasing fluencies of the picosecond laser to the optimal parameters in terms of efficacy and tolerance.

In a second phase, 10 additional subjects with black tattoos will be treated after central randomization on half of the tattoo with the picosecond laser (with the parameters determined in the first phase) and the other half treated with a nanosecond laser.

ELIGIBILITY:
Inclusion Criteria:

* Black tattoos with surface between 10 and 100 cm²
* Skin type I to VI

Exclusion Criteria:

* Childbearing age women
* Active dermatosis located on the tattoo
* Personal history of hypertrophic scars or keloids
* Pigmentary or vascular lesions located on the tattoo
* Subject taking oral steroid or retinoid or have any risk of delayed healing problems
* Acquired or hereditary conditions that could leead to a delayed healing
* Allergy to xylocaine, prilocaine or lidocaine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Percentage of decrease of tattoos 2 months after the third session as compared to baseline on standardized pictures | 2 month after the end of laser utilisation

SECONDARY OUTCOMES:
Evaluation of Pain with EVA test | 2 months after one session of laser utilisation
Evaluation of tolerance | 2 months after one session of laser utilisation
  correlation between EVA test and dermatological clinical signs
satisfaction evaluation of depigmanetation tattoo | 2 months after one session of laser utilisation
  satisfaction tests
Skin biopsies | immediately after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice - Dermatologie - Hôpital Archet, Nice, France